CLINICAL TRIAL: NCT00329134
Title: Investigation of the Efficacy of Quinine Sulphate Administered Via Taste-Masked Pellets to Children With Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Jean Paul Remon, University Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/177
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of quinine sulphate taste-masked pellets

SUMMARY:
No pediatric formulations of quinine exist. Therefore, quinine tablets are broken into 2 or 4 parts, according to the body weight. Based on the body weight, 1/2 or 1/4 a tablet is administered to the child.

At this moment, quinine sulphate pellets are developed. These pellets enable an adequate dosing according to the body weight.

56 children with malaria will be dosed every 8 hours during 7 days with 10-15mg/kg body weight.

ELIGIBILITY:
Inclusion Criteria:

* Malaria (falciparium malaria, uncomplicated)
* Informed consent

Exclusion Criteria:

-

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Clocktime when child has had no fever for minimal 48h (< 37,5°C)
Parasitemy

SECONDARY OUTCOMES:
Plasma concentration of quinine at day 4 between first and second administration

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Bortel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Centre Hospitalier De Butare, Butare, Rwanda

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be